CLINICAL TRIAL: NCT05390281
Title: Association Between Preoperative Level of Hemoglobin A1c and the Incidence of Acute Kindey Injury After Coronary Artery Bypass Grafting Surgery: a Cohort Study
Brief Title: Preoperative Level of Hemoglobin A1c and Acute Kindey Injury After Coronary Artery Bypass Grafting Surgery
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ghada M.Samir, Assistant Professor, Ain Shams University
Other Study IDs: FMASU MD 368/2018
Record Dates: First submitted 2022-05-14; First posted 2022-05-25 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Pre-diabetic group: Patients with preoperative HbA1c 5.7-6.4% (group A) (prediabetics)
  Interventions: Diagnostic Test: increase in serum creatinine
- Diabetic group: Patients with preoperative HbA1c > or = 6.5% till 7% or > 7% in case of emergency surgery or rapidly progressive cases with no time for long-term glycemic control (group B) (diabetics)
  Interventions: Diagnostic Test: increase in serum creatinine

INTERVENTIONS:
Diagnostic Test: increase in serum creatinine — any of the following: increase in serum creatinine by ≥ 0.3 mg/dl within 48 h of surgery or increase in serum creatinin

SUMMARY:
Background: The development of acute kidney injury (AKI) is an important indicator of clinical outcomes after cardiac surgery. Elevated preoperative hemoglobin A1c level may be associated with acute kidney injury in patients undergoing coronary artery bypass grafting. This study will investigate the association of preoperative HbA1c levels with AKI after isolated coronary artery bypass grafting (CABG).

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status II-III
* scheduled to undergo isolated coronary artery bypass grafting

Exclusion Criteria:

* Patients with history of renal failure
* Patients with history of hepatic failure
* Patients with history of heart failure
* previous cardiac surgery
* cerebrovascular event in the last 30 days
* percutaneous coronary intervention in the last 30 days prior to operation
* peripheral arterial disease
* malignancy
* infectious diseases
* patients who required surgical revision
* patients who required postoperative intra-aortic balloon pump
* patients with CBP time > 120 min or aortic cross clamp time > 90 min

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study compared the AKI incidence between patients with prediabetic level of HbA1c (5.7-6.4) and patients with elevated levels of HbA1c (> or = 6.5). Forty patients who underwent elective CABG were enrolled in this cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
serum creatinine level | 3 days
  increase in serum creatinine by ≥ 0.3 mg/dl within 48 h of surgery or increase in serum creatinine to ≥ 1.5 times baseline within 3 days of cardiac surgery

SECONDARY OUTCOMES:
Patients in need of RRT | 7 days
  The number of patients requiring postoperative renal replacement therapy

OTHER OUTCOMES:
Length of ICU stay | 7days
  The duration of postoperative patient stay in the intensive care

CONTACTS AND LOCATIONS:
Locations (1):
- Ain-Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No